CLINICAL TRIAL: NCT06018961
Title: Study of Postoperative Ileus in Digestive Surgery
Acronym: IPCID
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0491; 2022-A02834-39 (Other: ID-RCB)
Record Dates: First submitted 2023-07-18; First posted 2023-08-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Surgery
Keywords: Ileus; Colorectal surgery
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with digestive surgery: Patients who have planned abdominal surgery
  Interventions: Other: Post-operative ileus surgery

INTERVENTIONS:
Other: Post-operative ileus surgery — Collection of ileus events, items of IFEED score and surgical complications

SUMMARY:
Post-operative ileus is a temporary stoppage of bowel function following surgery. Indeed it can occur in 20% of cases during post-operative follow-up of bowel surgery. The absence of resumption of transit can lead to the implementation of specific treatments such as the placement of a nasogastric tube and drug treatments. To date, the definition of this event is not accepted by everyone and is not based on reproducible evaluation criteria. The main objective of this study is to evaluate a score used to date to define postoperative ileus, the IFEED score, and to compare it to the length of postoperative stay.

DETAILED DESCRIPTION:
Postoperative ileus (also known as paralytic ileus) is defined as a temporary cessation of gastrointestinal peristalsis. This complication occurs mainly following gastrointestinal surgery. It can be noted that postoperative ileus also occurs postoperatively after pelvic and extra-abdominal surgery with a lower incidence. The incidence of ileus varies depending on the cohorts, however the rate of occurrence can be up to 20% post-operative colorectal surgery.The main principles of treatment are the fasting of the patient and the introduction of a nasogastric tube to ensure gastric emptying in order to prevent complications of vomiting such as bronchial aspiration. This pathological phenomenon is frequent and significantly lengthens the duration of hospitalization and postoperative morbidity and mortality. The duration of hospitalization is the only objective and reproducible criterion in the evaluation of ileus. One of the problems of postoperative ileus is first of all its evaluation and the implementation of a reproducible definition. A recent consensus conference of the American Society for Engaged Recovery and Perioperative Quality Initiative proposed a return definition of transit based on an IFEED (Intake-Feeling Nauseated-Emesis-Physical Exam-Duration of Symptoms) clinical score. However, this score has never been evaluated prospectively in a cohort of patients operated on for pathologies of the digestive tract. This is a descriptive, diagnostic, prospective, monocentric study. We will include patients entering our care sector for a gastrointestinal surgery. We will follow patient from the surgery to the end of their hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patient entering our care sector for surgical management of a pathology affecting the digestive tract:
* Colorectal cancer
* Chronic inflammatory bowel disease
* Colonic diverticulosis.

Exclusion Criteria:

* Patient treated for digestive resection with associated resection procedure or to be treated with intraperitoneal chemotherapy.
* Patient presenting during hospitalization with an ileus secondary to another intra-abdominal complication.
* Patient cared for in an emergency
* Hepatic resection or other associated metastatic site
* Multiple digestive resection
* Colorectal anastomosis less than 7 cm from the anal margin (below the Pouch of Douglas)
* Patient with American Society of Anesthesiologists physical status (ASA) score > 2
* Patient with an Eastern Cooperative Oncology Group (ECOG) Performance Status Scale >2
* Pregnant or breastfeeding women
* Patient under a protection regime for adults (guardianship, curators, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population who have planned abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Complications of post-operative ileus surgery | 1 month
  Correlation between length of stay and Intake-Feeling nauseated-Emesis-physical Exam-Duration of symptoms (IFEED) score.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LE COSQUER, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHU de Toulouse, Toulouse
  - INSERM, Toulouse